CLINICAL TRIAL: NCT04110457
Title: Outcomes of Surgical Treatment of Patients With Spinal Metastasis in Assiut University Hospitals
Brief Title: Outcomes of Surgical Treatment of Patients With Spinal Metastasis in AUH
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim gamal asem, Principal investigator, Assiut University
Other Study IDs: surgical treatment in spine
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Spinal Metastases
MeSH Terms: interventions — Laminectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spinal decompression — spinal surgery by decompression or fixation

SUMMARY:
To analyze the outcomes of surgical treatment of patients with spinal metastases in spine unit in AUH regarding the pain control, neurological status and ambulatory status as well as survival rate .

DETAILED DESCRIPTION:
this study monitor what is the results after operative treatment of patients which have secondary metastases in spinal column concerning quality of live for one year and pain and neurology

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patient with tissue proven dx of cancer

Exclusion Criteria:

* Patient younger 18 years old
* CNS or spinal 1ry tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with spinal metastases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate quality of life after surgery | baseline
  to evaluate the general condition using 5Q-ED score

SECONDARY OUTCOMES:
to analyze postoperative pain control , stability and ambulatory statues after surgical treatment of spinal metastases. | Baseline
  evaluation of postoperative pain and neurology and comparing with preoperative data

CONTACTS AND LOCATIONS:
Overall Officials: Essam El morshidy, PHD, Study Director — lecturer
Locations (1):
- Assuit university, Asyut, Egypt

REFERENCES:
- [Background] Hirabayashi H, Ebara S, Kinoshita T, Yuzawa Y, Nakamura I, Takahashi J, Kamimura M, Ohtsuka K, Takaoka K. Clinical outcome and survival after palliative surgery for spinal metastases: palliative surgery in spinal metastases. Cancer. 2003 Jan 15;97(2):476-84. doi: 10.1002/cncr.11039. PMID 12518372
- [Result] Maccauro G, Spinelli MS, Mauro S, Perisano C, Graci C, Rosa MA. Physiopathology of spine metastasis. Int J Surg Oncol. 2011;2011:107969. doi: 10.1155/2011/107969. Epub 2011 Aug 10. PMID 22312491